CLINICAL TRIAL: NCT03754127
Title: A Comparative, Randomized Trial on HD-tDCS and Sham Control Group: Effects on Tinnitus Severity and Cognition Including Objective Measures.
Brief Title: A Randomized Controlled HD-tDCS Trial: Effects on Tinnitus Severity and Cognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Universiteit Antwerpen (Other)
Responsible Party: Principal Investigator, ethisch.comite@uza.be, Prof dr Annick Gilles (PhD), principal investigator, University Hospital, Antwerp
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EC 18/33/365
Record Dates: First submitted 2018-11-22; First posted 2018-11-27 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Tinnitus
Keywords: tinnitus; tdcs; neuromodulation; RCT
MeSH Terms: conditions — Tinnitus | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active group (Experimental): tDCS
  Interventions: Device: tDCS
- Sham group (Sham Comparator): Sham tDCS
  Interventions: Device: sham tDCS

INTERVENTIONS:
Device: tDCS — Transcranial direct current stimulation
  Arms: Active group
Device: sham tDCS — Sham transcranial direct current stimulation
  Arms: Sham group

SUMMARY:
This randomized, placebo-controlled study will compare the effects of HD-tDCS (a non-invasive neuromodulation technique) with a sham stimulation. In the sham situation, patients will undergo an identical treatment but no stimulation will be applied, allowing to control for placebo effects. This study will assess the effects of HD-tDCS on chronic, non-pulsatile tinnitus in a reliable way, as confounding factors such as anxiety, depression, hearing impairment, tinnitus gradation, age, and sex will be controlled for. Ultimately, this study will result in final recommendations for a standardised protocol for the use of HD-tDCS in tinnitus patients. When accurate, individualised, and effective therapy is available for the patient, the total cost (both economical and personal) will decrease significantly. The investigation's findings will be relevant for all caretakers dealing with tinnitus patients (psychologists, psychiatrists, manual therapists, general practitioners, ENT specialists, audiologists, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Duration of tinnitus: > 6 months
* 24 < TFI score < 90
* HADS depression subscale < 12
* HADS anxiety subscale < 12
* Hyperacusis questionnaire < 40
* Dutch- or Flemish-speaking

Exclusion Criteria:

* Somatic tinnitus
* Pregnancy
* Active middle ear pathology
* Hearing implants
* Known tumors in the head/neck region
* Patients having already had any other tinnitus treatment within the last 2 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Tinnitus Functional Index | 3 months
  The Tinnitus Functional Index (TFI) is a self-reported questionnaire, consisting of 25 questions, assessing the impact of tinnitus on patients' daily lives. The patient answers each question on a Likert scale ranging from 0 to 10. Questions 1 and 3 are expressed in percentages, and the Likert scale ranges from 0% to 100% (they are transformed to a 0-10 scale). The total score is then calculated as the mean of all questions multiplied by 10 to express this as a number between 0 and 100. In addition to the total score, the score of eight subscales can be determined. The subscales are the following: intrusiveness, reduced sense of control, cognitive interference, sleep disturbance, auditory difficulties attributed to tinnitus, interference with relaxation, reduced quality of life and emotional distress. A decrease of 13 points on the scale is considered as a clinical relevant difference.

SECONDARY OUTCOMES:
Tinnitus Questionnaire (TQ) | 3 months
  The Dutch validated version of the TQ is used to differentiate between emotional and cognitive distress, auditory difficulties, and self-experienced intrusiveness caused by the tinnitus. The total score can range from 0 to 84, assigning a subject to a distress category: slight (score = 0 - 30, grade 1), moderate (score = 31 - 46, grade 2), severe (score = 47 - 59, grade 3) and very severe (score = 60 - 84, grade 4).
Speech, Spatial and Qualities of Hearing Scale-12 (SSQ-12) | 3 months
  The SSQ12 is a short form of the Speech, Spatial and Qualities of Hearing scale. It is developed for use in clinical research and rehabilitation settings to measure a range of hearing disabilities across several domains such as speech in noise, speech in quiet, localization, distance and movement, segregation and listening effort. Responders rate their ability to do or experience the situation described in each question by marking a 1-10 scale (1 = not at all, 10 = perfectly). Scores of all 12 questions are averaged to obtain a global SSQ-12 score.
Hospital Anxiety and Depression Scale (HADS) | 3 months
  To detect states of depression and anxiety the Hospital Anxiety and Depression Scale (HADS) is used. This self-assessment questionnaire consists of seven items in the subscale 'depression' and seven items in the subscale 'anxiety' and distinguishes clearly between both emotional disorders. The HADS serves as a screening tool for depression and anxiety. Scores of 7 or less on each subscale indicate non-cases. Scores of 8-10 are borderline abnormal (borderline case), while scores of 11-21 are abnormal (case).
Visual Analogue Scale (VAS) | 3 months
  The patient scores the mean and maximum loudness of their tinnitus on a scale of 0 (absence of tinnitus) to 10 (as loud as possible, cannot be any louder).
Hyperacusis Questionnaire (HQ) | 3 months
  The HQ is a 14-item questionnaire that surveys a patient's hypersensitivity to sound. The 14 questions assess three dimensions (attentional, social, and emotional). The answer categories are: "no" (score of 0 points), "yes, a little" (1 point), "yes, quite a lot" (2 points), and "yes, a lot" (3 points). A total score of 28 or more indicates clinically significant hyperacusis.
Health Utility Index (HUI23) | 3 months
  The Health Utilities Index (HUI) is a family of generic health profiles and preference-based systems for the purposes of measuring health status, reporting health-related quality-of-life (QOL), and producing utility scores. The HUI comprises a 15-item questionnaire. The resulting total health-related QOL score ranges from 0.00 (dead) to 1.00 (perfect health).
Big Five Inventory-2 (BFI2) | 3 months
  The BFI2 comprises 60 statements to which subjects can assign a score ranging from 1 ('Disagree strongly') to 5 ('Agree strongly'). Each question belongs to one of the following 'Big Five' personality domains: Extraversion, Agreeableness, Conscientiousness, Negative Emotionality, and Open-Mindedness. For each domain, scores can vary from 12 to 60.
Speech-in-quiet (SPIQ) and speech-in-noise (SPIN) understanding | 3 months
Repeatable Battery for the Assessment of Neuropsychological Status, adjusted to test Hearing impaired individuals (RBANS-H) | 3 months
Cortical Auditory Evoked Potentials (CAEP) | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Antwerp University Hospital, Antwerp, Edegem, Belgium

REFERENCES:
- [Derived] Cardon E, Van Rompaey V, Jacquemin L, Mertens G, Vermeersch H, Joossen I, Beyers J, Vanderveken OM, Van de Heyning P, Topsakal V, Gilles A. Sequential dual-site High-Definition transcranial Direct Current Stimulation (HD-tDCS) treatment in chronic subjective tinnitus: study protocol of a double-blind, randomized, placebo-controlled trial. Trials. 2019 Aug 1;20(1):471. doi: 10.1186/s13063-019-3594-y. PMID 31370873